CLINICAL TRIAL: NCT07083687
Title: A Phase 2, Multi-Center, Open-Label, Single-Arm Study to Evaluate the Efficacy and Safety of Lorlatinib in TKI naïve, Advanced ROS1-Positive Non-Small Cell Lung Cancer Patients With Brain Metastases
Brief Title: Lorlatinib in ROS1+ NSCLC With Brain Metastasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-2025KY34
Record Dates: First submitted 2025-06-27; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer (NSCLC)
Keywords: non-small cell lung cancer; ROS1; lorlatinib
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — lorlatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 100mg lorlatinib QD Orally (Experimental)
  Interventions: Drug: Lorlatinib 100 mg

INTERVENTIONS:
Drug: Lorlatinib 100 mg — After enrollment, patients will receive 100 mg of lorlatinib orally once daily until disease progression, unacceptable toxicity, or withdraw study .

SUMMARY:
The goal of this Phase II, multicenter, open-label, single-arm clinical trial is to evaluate the intracranial efficacy and safety of lorlatinib in adults with TKI-naïve, advanced ROS1-positive non-small cell lung cancer (NSCLC) and untreated brain metastases. The main questions it aims to answer are:

What is the intracranial efficacy (eg., objective response rate/PFS) assessed by revised RECIST v1.1?

How do exploratory biomarkers (e.g., ctDNA dynamics in plasma/CSF) correlate with lorlatinib resistance?

Participants will:

Receive lorlatinib 100 mg orally once daily until disease progression or unacceptable toxicity.

Undergo brain MRI/CT scans every 8 weeks (first 12 cycles) and every 16 weeks thereafter.

Provide blood samples for safety/biomarker analysis and optional CSF samples via lumbar puncture during scheduled visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old.
2. Histologically or cytologically confirmed diagnosis of ROS1+ NSCLC with brain metastases before the use of lorlatinib.
3. ROS1 rearrangement positive confirmed by IHC FISH, PCR, or next generation sequencing (NGS). Patients with other treatable gene mutations besides ROS1 need to submit for discussion with the study experts to determine eligibility.
4. Treatment naïve or one prior systemic treatment with platinum-based chemotherapy.
5. Imaging (MR/CT) confirmed untreated brain metastases before lorlatinib initiation;
6. Participants with asymptomatic brain metastases or currently unrequiring corticosteroid treatment, or on a stable or decreasing dose of ≤10 mg QD prednisone or equivalent can be enrolled.
7. According to RECIST 1.1, patients must have at least one at least one measurable intracranial target lesion with the long axis greater or equal to 5 mm at baseline.
8. Eastern Cooperative Oncology Group Performance (ECOG) score of 0-1.
9. The subject's expected survival time must be 12 weeks or longer.
10. Participants must have normal primary organ function and meet the following criteria during screening:

（1）No blood transfusions within the past 14 days and Adequate hematopoietic function, defined as follows:

a） Hemoglobin > 90g/L（without the use of erythropoietin within the past 14 days） b） Absolute Neutrophil Count (ANC) ≥1.5×109/L（without the use of growth factors within the past 14 days） c） Platelets（PLT）≥100×109/L（without the use of platelet-stimulating agents within the past 14 days） （2）Adequate Liver Function, defined as follows：

1. Total serum bilirubin ≤1.5 x upper limit of normal (ULN)
2. Alanine Aminotransferase（ALT） and Aspartate Aminotransferase（AST）≤3.0 x ULN (≤5.0 x ULN in case of liver metastases) （3）Adequate Renal Function, defined as follows：

a） Serum creatinine（Cr）≤1.5× ULN or estimated creatinine clearance（CCr）≥45 ml/min （4）Adequate coagulation function, defined as follows：

a） International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN; PT can be within the predetermined range for the anticoagulant if the participant is currently receiving anticoagulant therapy Adequate Pancreatic Function, defined as serum total amylase≤1.5×ULN； 11.Adequate Pancreatic Function, defined as serum total amylase≤1.5×ULN； For women of childbearing potential (defined as not being postmenopausal for at least 1 year, or having undergone surgical sterilization or hysterectomy), a serum pregnancy test should be conducted within seven days prior to the first administration of the investigational drug, and the result should be negative. All participants (regardless of gender) must agree to use contraceptive measures during the entire treatment period and for at least 90 days after the last dose of the investigational drug.

12.Participants must understand and voluntarily sign the written informed consent form, demonstrate good compliance, adhere to the trial treatment plan and visit schedule, and be able to cooperate in observing adverse events and treatment efficacy.

Exclusion Criteria:

1. Have received treatment with the investigational drug or known allergy to the ingredients or excipients of the investigational drug.
2. Concurrent participation in another clinical study, except for observational (non-interventional) clinical studies or subsequent stages of interventional studies.
3. Brain metastasis combined with leptomeningeal metastases.
4. Brain metastasis with bleeding, or the presence of central nervous system complications requiring urgent local intervention (such as surgery, radiotherapy, etc.).
5. Presence of spinal cord compression unless pain symptoms and neurological function have remained stable or improved 2 weeks prior to enrollment.
6. Received open surgery (except surgery for biopsy purposes) within ≤14 days prior to enrollment.
7. Received intracranial radiotherapy before enrollment.
8. Fever with a temperature above 38℃ within the past week; or clinically significant bacterial, fungal, or viral infection, including but not limited to HIV infection, active HCV infection, active tuberculosis, active hepatitis B (active hepatitis B is defined as HBsAg positive and HBV-DNA copy number exceeds the upper limit of normal in the laboratory of the study center); or infections requiring hospitalization, septicemia, severe pneumonia, etc.
9. Significant clinical abnormalities in rhythm, conduction, or morphology on resting ECG, such as QT interval (QTc) ≥ 450 ms in males or ≥ 470 ms in females, complete left bundle branch block, 2nd degree or higher heart block, clinically significant ventricular arrhythmia, or atrial fibrillation.
10. Unstable angina, congestive heart failure (NYHA class III or IV), myocardial infarction, coronary/peripheral artery bypass, cerebrovascular accident, untreated transient ischemic attack, or symptomatic pulmonary embolism occurring currently or within the past 3 months.
11. Presence of risk factors for QT interval prolongation or increased risk of arrhythmia, such as grade 2 hypokalemia (grade 2 hypokalemia is defined as: blood potassium < normal lower limit -3.0mmol/L, and with symptoms, requiring treatment), congenital long QT syndrome, family history of long QT syndrome.
12. Past or current clinically active interstitial lung disease; presence of pulmonary interstitial fibrosis or active tuberculosis.
13. Disorders of swallowing function, active gastrointestinal disease, or other diseases significantly affecting the absorption, distribution, metabolism, and excretion of the investigational drug. History of major gastric resection.
14. Presence of other acquired, congenital immunodeficiency diseases, or previous solid organ or hematopoietic stem cell transplantation.
15. Evidence of severe or uncontrolled systemic diseases (such as severe mental, neurological diseases, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver or kidney diseases, uncontrolled hypertension i.e., still being greater than or equal to CTCAE 5.0 grade 3 hypertension after drug treatment).
16. Diagnosis or treatment of other malignant tumors within the past 5 years (excluding adequately treated basal cell or squamous cell skin cancer, bladder carcinoma in situ, cervical carcinoma in situ, ductal carcinoma in situ, localized prostate cancer).
17. Use of any known QT-prolonging drugs within 2 weeks before the first dose.
18. Use or consumption of known potent CYP3A4 inhibitors in medications or food within the past 2 weeks; use of known potent CYP3A4 inducers within the past 2 weeks; use of medications that act as CYP3A4 substrates (with a narrow therapeutic index) within the past 2 weeks.
19. Severe acute or chronic mental illness, including recent (within the past year) or active suicidal ideation or behavior.
20. For pregnant or lactating women or male or female participants with reproductive potential, refusal to adopt effective contraceptive measures during the treatment period and for 90 days after the last use of the investigational drug.
21. The investigator believes that the participant may be unable to complete the study or comply with the study requirements.
22. The investigator believes that there are other potential risks making the participant unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial Objective Response Rate (iORR), based on the modified version 1.1 of the Response Evaluation Criteria in Solid Tumors (RECIST) | up to 26 weeks

IPD SHARING:
Plan to Share IPD: Undecided